CLINICAL TRIAL: NCT03781778
Title: Randomized, Controlled Trial of Resistant Starch in Stage I-Ill Colorectal Cancer Survivors Pilot Study: The Fiber for Health After Cancer Study
Brief Title: Pilot Trial of Resistant Starch in Stage I-III Colorectal Cancer Survivors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to expiration of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marian Neuhouser, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1003387; NCI-2018-02802 (Other: NCI / CTRP); 10079 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Colon Cancer; Rectal Cancer; Cancer Survivor; Colorectal Adenocarcinoma; Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8
Keywords: Resistant Starch; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Diet Therapy; Resistant Starch

STUDY DESIGN:
Intervention Model Description: Blinded, block randomization based on sex and BMI.
Who Masked: Participant, Investigator
Masking Description: Assignment to the active versus control group will be blinded using a computer program and will be designated as "diet A" and "diet B". Investigators will be unblinded once the study and data analyses have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (resistant starch foods) (Experimental): Patients eat a diet consisting of resistant starch foods daily for 8 weeks.
  Interventions: Other: Dietary Intervention (resistant starch); Other: Questionnaire Administration
- Group II (foods with regular corn starch) (Active Comparator): Patients eat a diet consisting of regular corn starch foods daily for 8 weeks.
  Interventions: Other: Dietary Intervention (regular starch); Other: Questionnaire Administration

INTERVENTIONS:
Other: Dietary Intervention (resistant starch) — Eat foods with resistant starch
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Group I (resistant starch foods)
Other: Dietary Intervention (regular starch) — Eat foods with regular corn starch
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Group II (foods with regular corn starch)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II, randomized pilot trial studies the effect of the consumption of foods made with resistant starch compared to foods made with corn starch on biomarkers that may be related to colorectal cancer progression in stage I-III colorectal cancer survivors. Foods made with resistant starch may beneficially influence markers of inflammation, insulin resistance, and the composition of gut bacteria in colorectal cancer survivors.

DETAILED DESCRIPTION:
Participants are randomized to 1 of 2 groups.

GROUP I (INTERVENTION GROUP): Participants eat a diet consisting of resistant starch foods daily for 8 weeks. Study provided foods are in addition to their own usual daily diet.

GROUP II (CONTROL GROUP): Participants eat a diet consisting of regular corn starch foods daily for 8 weeks. Study provided foods are in addition to their own usual daily diet.

ELIGIBILITY:
Inclusion Criteria:

* History of diagnosed American Joint Committee on Cancer (AJCC) stage I-III colorectal adenocarcinoma.
* Completed all treatment of colorectal adenocarcinoma within past 4-36 months.
* Current Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (per physician).
* Ability to consent and follow study protocol.

Exclusion Criteria:

* Active cancer.
* Prior diagnosis of diabetes that is currently uncontrolled (defined as hemoglobin [Hgb] A1c > 8.0).
* Active inflammatory bowel disease (i.e., patients who are symptomatic despite medical therapy). This includes irritable bowel syndrome, Crohn's disease, or any other inflammatory bowel disorder.
* Known food allergy/intolerances to wheat, gluten, dairy or eggs.
* Use of antibiotic(s) within the last 3 months prior to enrollment.
* Women who are pregnant and/or breastfeeding.
* Current body mass index (BMI) < 18.5 kg/m^2.
* Uncontrolled constipation.
* Inability to speak and fully understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Neuhouser, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-Active (Resistant Starch): Participants receive daily study snack foods prepared with resistant starch. Dosing is 15g of starch daily for the first 14 days, then 30g of starch daily for the remaining 42 days.
- 2-Control (Regular Starch): Participants receive daily study snack foods prepared with regular starch. Dosing is 15g of starch daily for the first 14 days, then 30g of starch daily for the remaining 42 days.
Period: Overall Study
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Started | 4 | 6
Started Intervention | 3 | 4
Completed | 2 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: at time of enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch) | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [55 to 68] | 50 [38 to 79] | 58.5 [38 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10
Height [Median (Full Range); unit: cm] | 177.54 [168.00 to 180.10] | 173.75 [156.21 to 187.00] | 176.00 [156.21 to 187.00]
Weight [Median (Full Range); unit: kg] | 85.88 [67.90 to 96.16] | 88.95 [50.58 to 113.10] | 85.90 [50.58 to 113.10]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 27.7 [21.2 to 32.7] | 27.2 [20.7 to 38.5] | 27.65 [20.7 to 38.5]
BMI Category [Count of Participants; unit: Participants]
  Underweight | 0 | 0 | 0
  Normal weight | 1 | 3 | 4
  Overweight | 2 | 0 | 2
  Obese I | 1 | 2 | 3
  Obese II+ | 0 | 1 | 1
T-stage [Count of Participants; unit: Participants] — Participants were staged clinically by the interdisciplinary clinical oncology team per American Joint Committee on Cancer Staging Criteria for colorectal carcinoma (AJCC 8th edition). AJCC Stage Groupings I-III for colorectal carcinoma were eligible for the trial. Prognostic outcomes are considered better for lower stages and worse for higher stages.
  Participants
    T0 | 0 | 0 | 0
    T1 | 0 | 0 | 0
    T2 | 0 | 1 | 1
    T3 | 3 | 5 | 8
    T4a | 1 | 0 | 1
    T4b | 0 | 0 | 0
N-stage [Count of Participants; unit: Participants] — Participants were staged clinically by the interdisciplinary clinical oncology team per American Joint Committee on Cancer Staging Criteria for colorectal carcinoma (AJCC 8th edition). AJCC Stage Groupings I-III for colorectal carcinoma were eligible for the trial. Prognostic outcomes are considered better for lower stages and worse for higher stages.
  Participants
    N0 | 0 | 2 | 2
    N1 | 1 | 0 | 1
    N1a | 1 | 1 | 2
    N1b | 0 | 1 | 1
    N1c | 1 | 2 | 3
    N2 | 1 | 0 | 1
    N2a | 0 | 0 | 0
    N2b | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Accrual
Description: The accrual rate will be estimated with number of participants at full enrollment at 12 months.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 4 | 5
Participants | 4 | 5

2. Primary Outcome: Feasibility: Adherence
Description: The adherence endpoint pertains to adherence to the intervention and is defined as consuming 75% or more of study foods on 75% of days from baseline to 8 weeks.
Time Frame: From start of intervention to ending intervention: up to 8 weeks
Population: Overall number of participants analyzed for the adherence measure: 7 (per protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 3 | 4
Participants | 2 | 4

3. Primary Outcome: Feasibility: Retention
Description: The retention endpoint is defined as at least 80% of enrolled participants providing blood and stool samples at the week 8 timepoint.
Time Frame: From start of intervention to the 8-week timepoint
Population: All participants enrolled, in accordance with protocol and Statistical Analysis Plan
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 4 | 6
Participants | 3 | 5

4. Secondary Outcome: Variability of Biomarkers of Insulin Resistance and Inflammation (Adiponectin)
Description: Adiponectin was measured at baseline and week 8 (follow-up) and reported using descriptive statistics.
Time Frame: Baseline to follow-up at week 8
Population: Of the 10 participants enrolled to the study, blood was collected at the baseline and week 8 follow-up timepoints on just 5 participants.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 2 | 3
ug/mL
  Adiponectin - baseline | 1.33 (0.54) | 1.95 (0.95)
  Adiponectin - followup | 1.14 (0.55) | 2.08 (1.11)

5. Secondary Outcome: Variability in Biomarkers of Insulin Resistance and Inflammation (C-reactive Protein, CRP)
Description: CRP was measured at baseline and week 8 (follow-up) and reported using descriptive statistics.
Time Frame: Baseline to follow-up at week 8
Population: Of the 10 participants enrolled to the study, blood was collected at the baseline and week 8 followup timepoints on just 5 participants.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 2 | 3
mg/L
  C-reactive protein - baseline | 1.24 (0.74) | 1.98 (2.13)
  C-reactive protein - followup | 1.93 (2.37) | 1.67 (1.77)

6. Secondary Outcome: Variability in Gut Microbial Communities From Human Stool Samples - ALPHA DIVERSITY AND GENERA
Description: This measure assesses variability in gut microbial communities from human stool samples collected during the study by changes in alpha diversity and genera in response to the intervention. We will use multivariate and univeriate approaches to assess significant changes int he microbiome in response to the intervention.
Time Frame: Baseline to follow-up at weeks 2 and 8
Population: Of the 10 participants enrolled to this study, fecal samples were collected at baseline and followup for 7 participants. Of these 7 participants, one participant on Arm 1 dropped out of the study after week 2 hence the week 8 followup fecal was not obtained. For the remaining 6 participants, fecal samples from all three time-points were analyzed.
Measure: Mean (Standard Deviation); unit: Relative abundance
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 3 | 4
Relative abundance
  Alpha diversity - baseline | 1344 (243.50) | 1458 (265.20)
  Alpha diversity - first follow-up (week 2) | 1376 (21.70) | 1111 (364.00)
  Alpha diversity - second follow-up (week 8) | 1288 (2.83) | 1321 (75.40)
  Faecalibacterium Prausnitzii - baseline | 2.09 (1.31) | 2.62 (2.52)
  Faecalibacterium Prausnitzii - first follow-up (week 2) | 1.84 (1.02) | 1.77 (2.12)
  Faecalibacterium Prausnitzii - second follow-up (week 8) | 0.98 (0.52) | 2.09 (1.73)
  Akkermansia mucinipiila - baseline | 0.36 (0.22) | 0.35 (0.29)
  Akkermansia mucinipiila - first follow-up (week 2) | 0.19 (0.05) | 0.18 (0.11)
  Akkermansia mucinipiila - second follow-up (week 8) | 0.19 (0.02) | 0.39 (0.48)

7. Secondary Outcome: Variability in Gut Microbial Communities From Human Stool Samples -- BETA DIVERSITY
Description: This measure assesses variability in gut microbial communities from human stool samples collected during the study by changes in global microbial community (beta diversity) in response to the intervention. We will use multivariate and univeriate approaches to assess significant changes in the microbiome in response to the intervention.
Time Frame: Baseline to followup at weeks 2 and 8
Population: Analysis limitation: due to low participant recruitment, there was insufficient number of stool samples available to detect and compute beta diversity.
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of intervention to ending the intervention: up to 8 weeks.
Description: Method of assessment: weekly participant-completed questionnaire. The number of participants (n=7) analyzed for adverse events ("number at risk" below) is fewer than the number enrolled (n=10) because 3 participants withdrew consent prior to starting the intervention.
Arm/Group | 1-Active (Resistant Starch) | 2-Control (Regular Starch)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Active (Resistant Starch) (N=3) | 2-Control (Regular Starch) (N=4)
Gassiness (Gastrointestinal disorders) | 2 (2) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1) | 3 (3)
Increased frequency of bowel movements (Gastrointestinal disorders) | 1 (1) | 2 (2)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose stool (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03781778/Prot_SAP_000.pdf